CLINICAL TRIAL: NCT04919772
Title: Assessing the Reliability and Validity of 4-meter and 10-meter Walking Test for Measurements of Gait Speed and Their Correlation With 5-repetition Sit-to-stand Test in Chronic Stroke Survivors
Brief Title: Assessing the Reliability and Validity of 4-meter and 10-meter Walking Test
Status: Completed | Type: Observational
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, Rosa Cabanas Valdés, Principal investigator, Universitat Internacional de Catalunya
Other Study IDs: 4-meter walking test
Record Dates: First submitted 2021-05-23; First posted 2021-06-09 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Stroke; Gait, Hemiplegic; Cerebral Infarction; Cerebrovascular Disorders
Keywords: walking speed; gait; sit-to-stand; reliability; validity; correlation
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic; Cerebral Infarction; Cerebrovascular Disorders | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke survivors: Chronic stroke, generally speaking chronic stroke refers to the period of recovery that takes place at least six months after the initial stroke event
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — The participants walk 4-meter and 10-meter and 5-repetition sit-to-stand twice.
  Other Names: Evaluation

SUMMARY:
The 4-meter walk test and 10-meter walk test is currently applied to assess gait speed.These tools are frequently used in clinical trials and were also shown to be reliable measurement methods. There are ocassions where it is not possible to have a long corridor to measure gait speed. It is necessary to have a tool to evaluate gait speed in a small space as 4-meter walk test.

DETAILED DESCRIPTION:
Walking speed is an important aspect of gait and is commonly used as an objective measure of functional mobility in both clinical and research settings. The majority who have suffered a stroke tend to have gait disturbances. Regaining locomotor ability is one of the primary goals in stroke rehabilitation, and it is most commonly measured using changes in self-selected walking speed. Although many of them can walk independently, they do not do so with enough speed and endurance to allow them to perform their activities of daily living prior to stroke. Not only is self-selected walking speed simple, cost effective, reliable, valid, sensitive, and specific, but it is also highly related to the severity of impairment and predicts functional walking status. It is recommended as a "vital sign" of health. Improvements in walking speed of 0.1 m/s or more have been shown to be a predictor of good health. However, decreased walking speed has been related to worse health outcomes and frailty in older people.

The 4-meter walk test (4 MWT) and 10-meter walk test (10 MWT) is currently applied using various timing protocols and distance covered that may affect data interpretation with a standard value, and comparisons among the studies. There are two protocols to measure walking speed, static and flying start. A static start (i.e., record the time used to cover a total walkway or from the start to stop walking) or a flying start (i.e., measured the time while walking in the middle of the walkway).

The aim of this study is to investigate the test-retest reliability of the 4 MWT and 10 MWT and their correlation with 5-repetition sit-to-stand in chronic stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* All study participants are clinically diagnosed with stroke
* Adult participants, defined as >18 years of age
* Have preserved cognitive ability: Achieve a score equal to or greater than 25 points on the Montreal Cognitive Assessment test.
* Have the ability to walk on a flat surface of at least 20 meters, with or without aid.

Exclusion Criteria:

* A history of lower extremities injury or surgery
* A history of botulinum injection within 3 months
* A history of inflammatory arthritis
* A history of inflammatory myopathy or peripheral nervous disease
* A history of other neurological disease as a Parkinson, spinal cord etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke survivors in chronic phase > 6 months
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Reliability of 4-meter walking test | Baseline
  Reliability is the overall consistency of a measure.
Reliability of 4-meter walking test | 1 hour later from baseline
  Reliability is the overall consistency of a measure.
Validity of 4-meter walking test | Baseline
  Validity is the extent to which a concept, conclusion or measurement is well-founded and likely corresponds accurately to the real world
Validity of 4-meter walking test | 1 hour later from baseline
  Validity is the extent to which a concept, conclusion or measurement is well-founded and likely corresponds accurately to the real world
Reliability of 10-meter walking test | Baseline
  Reliability is the overall consistency of a measure.
Reliability of 10-meter walking test | 1 hour later from baseline
  Reliability is the overall consistency of a measure.
Validity of 10-meter walking test | Baseline
  Validity is the extent to which a concept, conclusion or measurement is well-founded and likely corresponds accurately to the real world
Validity of 10-meter walking test | 1 hour later from baseline
  Validity is the extent to which a concept, conclusion or measurement is well-founded and likely corresponds accurately to the real world

SECONDARY OUTCOMES:
Correlation of 5-repetition sit-to-stand with 4-meter walking test | Baseline
  A rank correlation coefficient measures the degree of similarity between two rankings, and can be used to assess the significance of the relation between them.
Correlation of 5-repetition sit-to-stand with 10-meter walking test | Baseline
  A rank correlation coefficient measures the degree of similarity between two rankings, and can be used to assess the significance of the relation between them.

CONTACTS AND LOCATIONS:
Overall Officials: Laura García-Rueda, MsC, Study Director — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Barcelona, Spain

REFERENCES:
- [Background] Bohannon RW. Measurement of gait speed of older adults is feasible and informative in a home-care setting. J Geriatr Phys Ther. 2009;32(1):22-3. doi: 10.1519/00139143-200932010-00005. PMID 19856632
- [Background] Karpman C, Lebrasseur NK, Depew ZS, Novotny PJ, Benzo RP. Measuring gait speed in the out-patient clinic: methodology and feasibility. Respir Care. 2014 Apr;59(4):531-7. doi: 10.4187/respcare.02688. Epub 2013 Aug 27. PMID 23983271
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Result] Richards CL, Malouin F, Dean C. Gait in stroke: assessment and rehabilitation. Clin Geriatr Med. 1999 Nov;15(4):833-55. PMID 10499938
- [Result] Eng JJ, Tang PF. Gait training strategies to optimize walking ability in people with stroke: a synthesis of the evidence. Expert Rev Neurother. 2007 Oct;7(10):1417-36. doi: 10.1586/14737175.7.10.1417. PMID 17939776
- [Result] Jorgensen HS, Nakayama H, Raaschou HO, Olsen TS. Recovery of walking function in stroke patients: the Copenhagen Stroke Study. Arch Phys Med Rehabil. 1995 Jan;76(1):27-32. doi: 10.1016/s0003-9993(95)80038-7. PMID 7811170
- [Result] Geyh S, Cieza A, Schouten J, Dickson H, Frommelt P, Omar Z, Kostanjsek N, Ring H, Stucki G. ICF Core Sets for stroke. J Rehabil Med. 2004 Jul;(44 Suppl):135-41. doi: 10.1080/16501960410016776. PMID 15370761
- [Result] Parker CJ, Gladman JR, Drummond AE. The role of leisure in stroke rehabilitation. Disabil Rehabil. 1997 Jan;19(1):1-5. doi: 10.3109/09638289709166438. PMID 9021278
- [Result] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Result] Awad L, Reisman D, Binder-Macleod S. Distance-Induced Changes in Walking Speed After Stroke: Relationship to Community Walking Activity. J Neurol Phys Ther. 2019 Oct;43(4):220-223. doi: 10.1097/NPT.0000000000000293. PMID 31449180
- [Result] Montero-Odasso M, Schapira M, Soriano ER, Varela M, Kaplan R, Camera LA, Mayorga LM. Gait velocity as a single predictor of adverse events in healthy seniors aged 75 years and older. J Gerontol A Biol Sci Med Sci. 2005 Oct;60(10):1304-9. doi: 10.1093/gerona/60.10.1304. PMID 16282564
- [Result] Feld JA, Rabadi MH, Blau AD, Jordan BD. Berg balance scale and outcome measures in acquired brain injury. Neurorehabil Neural Repair. 2001;15(3):239-44. doi: 10.1177/154596830101500312. PMID 11944746
- [Result] Taylor-Piliae RE, Latt LD, Hepworth JT, Coull BM. Predictors of gait velocity among community-dwelling stroke survivors. Gait Posture. 2012 Mar;35(3):395-9. doi: 10.1016/j.gaitpost.2011.10.358. Epub 2011 Nov 26. PMID 22119886
- [Result] Braden HJ, Hilgenberg S, Bohannon RW, Ko MS, Hasson S. Gait speed is limited but improves over the course of acute care physical therapy. J Geriatr Phys Ther. 2012 Jul-Sep;35(3):140-4. doi: 10.1519/JPT.0b013e31824baa1e. PMID 22415359
- [Result] Barthuly AM, Bohannon RW, Gorack W. Gait speed is a responsive measure of physical performance for patients undergoing short-term rehabilitation. Gait Posture. 2012 May;36(1):61-4. doi: 10.1016/j.gaitpost.2012.01.002. Epub 2012 Mar 8. PMID 22406292
- [Result] Hardy SE, Perera S, Roumani YF, Chandler JM, Studenski SA. Improvement in usual gait speed predicts better survival in older adults. J Am Geriatr Soc. 2007 Nov;55(11):1727-34. doi: 10.1111/j.1532-5415.2007.01413.x. Epub 2007 Oct 3. PMID 17916121
- [Result] Middleton A, Fritz SL, Lusardi M. Walking speed: the functional vital sign. J Aging Phys Act. 2015 Apr;23(2):314-22. doi: 10.1123/japa.2013-0236. Epub 2014 May 2. PMID 24812254
- [Result] Graham JE, Ostir GV, Fisher SR, Ottenbacher KJ. Assessing walking speed in clinical research: a systematic review. J Eval Clin Pract. 2008 Aug;14(4):552-62. doi: 10.1111/j.1365-2753.2007.00917.x. Epub 2008 May 2. PMID 18462283
- [Result] Amatachaya S PT, PhD, Kwanmongkolthong M PT, BSc, Thongjumroon A PT, BSc, Boonpew N PT, BSc, Amatachaya P ME, PhD, Saensook W PT PhD, Thaweewannakij T PT, PhD, Hunsawong T PT, PhD. Influence of timing protocols and distance covered on the outcomes of the 10-meter walk test. Physiother Theory Pract. 2020 Dec;36(12):1348-1353. doi: 10.1080/09593985.2019.1570577. Epub 2019 Feb 1. PMID 30704332
- [Result] Cheng DK, Nelson M, Brooks D, Salbach NM. Validation of stroke-specific protocols for the 10-meter walk test and 6-minute walk test conducted using 15-meter and 30-meter walkways. Top Stroke Rehabil. 2020 May;27(4):251-261. doi: 10.1080/10749357.2019.1691815. Epub 2019 Nov 21. PMID 31752634
- [Result] Wade DT, Hewer RL. Functional abilities after stroke: measurement, natural history and prognosis. J Neurol Neurosurg Psychiatry. 1987 Feb;50(2):177-82. doi: 10.1136/jnnp.50.2.177. PMID 3572432
- [Result] Unver B, Baris RH, Yuksel E, Cekmece S, Kalkan S, Karatosun V. Reliability of 4-meter and 10-meter walk tests after lower extremity surgery. Disabil Rehabil. 2017 Dec;39(25):2572-2576. doi: 10.1080/09638288.2016.1236153. Epub 2016 Oct 11. PMID 27728985
- [Result] Peters DM, Fritz SL, Krotish DE. Assessing the reliability and validity of a shorter walk test compared with the 10-Meter Walk Test for measurements of gait speed in healthy, older adults. J Geriatr Phys Ther. 2013 Jan-Mar;36(1):24-30. doi: 10.1519/JPT.0b013e318248e20d. PMID 22415358
- [Result] Mokkink LB, Terwee CB, Knol DL, Stratford PW, Alonso J, Patrick DL, Bouter LM, de Vet HC. Protocol of the COSMIN study: COnsensus-based Standards for the selection of health Measurement INstruments. BMC Med Res Methodol. 2006 Jan 24;6:2. doi: 10.1186/1471-2288-6-2. PMID 16433905
- [Derived] Cabanas-Valdes R, Garcia-Rueda L, Salgueiro C, Perez-Bellmunt A, Rodriguez-Sanz J, Lopez-de-Celis C. Assessment of the 4-meter walk test test-retest reliability and concurrent validity and its correlation with the five sit-to-stand test in chronic ambulatory stroke survivors. Gait Posture. 2023 Mar;101:8-13. doi: 10.1016/j.gaitpost.2023.01.014. Epub 2023 Jan 20. PMID 36696822